CLINICAL TRIAL: NCT01380899
Title: Usefulness of α-synuclein as a Marker for Early Diagnosis of Parkinson's Disease in Skin Biopsy.
Status: Completed | Type: Observational
Sponsor: Universidad Autonoma de San Luis Potosí (Other)
Responsible Party: Principal Investigator, Ildefonso Rodriguez-Leyva, MD, PhD, FAAN, FANA, Universidad Autonoma de San Luis Potosí
Other Study IDs: UASLP-PD001
Record Dates: First submitted 2011-06-17; First posted 2011-06-27 (Estimated); Results first posted 2021-05-25 (Actual); Last update posted 2021-05-25 (Actual); Status verified 2021-05

CONDITIONS: Parkinson Disease; Parkinsonian Disorders
Keywords: Parkinson Disease; Parkinsonian Disorders; Lewy Bodies; alpha-Synuclein
MeSH Terms: conditions — Parkinson Disease; Parkinsonian Disorders; Parkinson Disease 4, Autosomal Dominant Lewy Body

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — We are obtaining the skin of the participants, by biopsy using a punch 3-4 mm in retro auricular area.
  We are taking from affected subjects and his or her partner (the most husband or wife).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- PD Parkinson´s Disrease: We are studying the presence of alpha-synuclein in the epidermis and dermis besides the end nerve terminal. We have several reports until now, and we are following the study because we wish to convince the academic and scientific society over the utility of this study to be close to the molecular diagnosis of this kind of disease.
  Interventions: Procedure: Biopsy of skin
- AP Atypical Parkinsonism: with neurodegenerative disease (proteinopathies) and secondary AP.
- Control group: Subjects without neurodegenerative disease and apparently good health status with an age that matches the problems groups

INTERVENTIONS:
Procedure: Biopsy of skin — Under local anesthesia with 1% xylocaine, 4-mm punch biopsies with 3-mm depth, including the dermis and subcutaneous fat tissue, will undergone from two regions, neck and lower back.
  Groups: PD Parkinson´s Disrease

SUMMARY:
Parkinson's disease (PD) is a degenerative disease that can be difficult to diagnose. The clinicopathological studies had demonstrated a 76% accuracy in the clinical diagnosis of PD.

At the beginning of PD is difficult for the clinician to distinguish from Parkinsonism Plus Syndromes (PPS) due to the similarity of symptoms and the lack of specific diagnostic tests.

Specific biomarkers to help improve the accuracy of diagnosis and to separate these two entities are highly needed

The histological hallmark for definite diagnosis of PD is the presence of fibrillar aggregates of phosphorylated alpha-synuclein called Lewy bodies (LBs) and Lewy neurites. Previous autopsy-based studies have revealed that alpha-synuclein is deposited in the peripheral autonomic nervous system including the enteric nervous system of the alimentary tract, cardiac plexus, adrenal medulla and skin.

For this reason, in patients with parkinsonism, an alternative tool could be to demonstrate alpha-synuclein fibrillar aggregates in the skin, allowing early and appropriate diagnosis.

DETAILED DESCRIPTION:
Parkinsonism, the syndrome, is a common movement disorder, and Parkinson's disease, the most common cause of parkinsonism, is the second most prevalent neurodegenerative disease after Alzheimer's disease.

The clinical diagnosis of PD is based on the presence of the four common features: tremor when the limb is at rest, resistance to passive movement of the joints (rigidity), slowness and paucity of movement (bradykinesia and akinesia) and postural abnormalities.

Approximately 25 percent of patients who received an initial clinical diagnosis of PD are found to have parkinsonism as part of another disorder, such as one of the so-called Parkinsonism-Plus Syndromes (PPS) The number and complexity of PPS seem to be increasing. This, along with the lack of diagnostic tests, makes it difficult for the clinician to distinguish between disease types.

Some characteristic clinical features are used for the differential diagnosis, this manifestations include early and severe postural instability, falls in the first year of onset, abnormal eye movements, autonomic dysfunction, cerebellar signs and upper motor neuron signs. The PPS respond poorly to antiparkinsonian medications and have a worse prognosis than does PD. In spite of these suggestive features, not all PD patients have the same progression, in some cases it is impossible to separate typical PD from PPS, especially at the early stage. In this context, biological markers must be of great usefulness for the differential diagnosis of these entities.

Some reports have described early features of PD such as (SPECT) imaging of the dopamine transporter that demonstrated the reduction of dopamine transporter in the striatum body at the early stage of PD and degeneration of the cardiac sympathetic nerve at the beginning of the disease process of PD; this occurs before neuronal cell loss is present in the dorsal vagal nucleus; This fact accounts for reduced cardiac uptake of meta-iodobenzylguanidine (MIBG), a physiological analog of norepinephrine. However, these diagnostic methods are not often performed. Therefore, more sensitive methods are needed to help improve the accuracy of diagnosis of PD.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Parkinson's Disease or Parkinson Plus Syndrome
* Subject is a male or female between the age of 50 and 95
* Subject will write the informed consent

Exclusion Criteria:

* History of stroke or/and trauma
* Signs of cerebrovascular pathology
* Brain tumor
* Severe unrelated neurological or physical disease

Ages: 35 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The patients will be selected from the department of neurology and the office of the principal investigator.
Sampling Method: Non-Probability Sample
Enrollment: 87 (Actual)
Dates: Start 2011-02; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ildefonso Rodríguez-Leyva, MD, Principal Investigator — Hospital Central "Dr. Ignacio Morones Prieto"; Maria E Jimenez-Capdeville, PhD, Study Director — Universidad Autonoma de San Luis Potosi; Juan P Castanedo-Cazares, MD, Study Director — Hospital Dr. Ignacio Morones Prieto; Erika G Chi-Ahumada, MC, Study Chair — Facultad de Medicina, UASLP; Maria E Jimenez-Capdeville, PhD, Study Chair — Facultad de Medicina; Robert A. Norman, MD, PhD., Study Chair — Independent Dermatologist
Locations (1):
- Hospital Central Dr. Ignacio Morones Prieto, San Luis Potosí City, Mexico

IPD SHARING:
Plan to Share IPD: No
Each participant has to sign the concern form. We can share his clinical data, but not private information.

REFERENCES:
- [Background] Nutt JG, Wooten GF. Clinical practice. Diagnosis and initial management of Parkinson's disease. N Engl J Med. 2005 Sep 8;353(10):1021-7. doi: 10.1056/NEJMcp043908. No abstract available. PMID 16148287
- [Background] Gelb DJ, Oliver E, Gilman S. Diagnostic criteria for Parkinson disease. Arch Neurol. 1999 Jan;56(1):33-9. doi: 10.1001/archneur.56.1.33. PMID 9923759
- [Background] Hughes AJ, Daniel SE, Kilford L, Lees AJ. Accuracy of clinical diagnosis of idiopathic Parkinson's disease: a clinico-pathological study of 100 cases. J Neurol Neurosurg Psychiatry. 1992 Mar;55(3):181-4. doi: 10.1136/jnnp.55.3.181. PMID 1564476
- [Background] Tuite PJ, Krawczewski K. Parkinsonism: a review-of-systems approach to diagnosis. Semin Neurol. 2007 Apr;27(2):113-22. doi: 10.1055/s-2007-971174. PMID 17390256
- [Background] Ibanez-Salazar A, Banuelos-Hernandez B, Rodriguez-Leyva I, Chi-Ahumada E, Monreal-Escalante E, Jimenez-Capdeville ME, Rosales-Mendoza S. Oxidative Stress Modifies the Levels and Phosphorylation State of Tau Protein in Human Fibroblasts. Front Neurosci. 2017 Sep 7;11:495. doi: 10.3389/fnins.2017.00495. eCollection 2017. PMID 28936161
- [Result] Rodriguez-Leyva I, Calderon-Garciduenas AL, Jimenez-Capdeville ME, Renteria-Palomo AA, Hernandez-Rodriguez HG, Valdes-Rodriguez R, Fuentes-Ahumada C, Torres-Alvarez B, Sepulveda-Saavedra J, Soto-Dominguez A, Santoyo ME, Rodriguez-Moreno JI, Castanedo-Cazares JP. alpha-Synuclein inclusions in the skin of Parkinson's disease and parkinsonism. Ann Clin Transl Neurol. 2014 Jul;1(7):471-8. doi: 10.1002/acn3.78. Epub 2014 Jul 1. PMID 25356418
- [Result] Rodriguez-Leyva I, Chi-Ahumada EG, Carrizales J, Rodriguez-Violante M, Velazquez-Osuna S, Medina-Mier V, Martel-Gallegos MG, Zarazua S, Enriquez-Macias L, Castro A, Calderon-Garciduenas AL, Jimenez-Capdeville ME. Parkinson disease and progressive supranuclear palsy: protein expression in skin. Ann Clin Transl Neurol. 2016 Feb 1;3(3):191-9. doi: 10.1002/acn3.285. eCollection 2016 Mar. PMID 27042679
- [Result] Rodriguez-Leyva I, Chi-Ahumada E, Mejia M, Castanedo-Cazares JP, Eng W, Saikaly SK, Carrizales J, Levine TD, Norman RA, Jimenez-Capdeville ME. The Presence of Alpha-Synuclein in Skin from Melanoma and Patients with Parkinson's Disease. Mov Disord Clin Pract. 2017 Jun 1;4(5):724-732. doi: 10.1002/mdc3.12494. eCollection 2017 Sep-Oct. PMID 30363411
- [Result] Mejia M, Rodriguez-Leyva I, Cortes-Enriquez F, Chi-Ahumada E, Portales-Perez DP, Macias-Islas MA, Jimenez-Capdeville ME. Low levels of alpha-synuclein in peripheral tissues are related to clinical relapse in relapsing-remitting multiple sclerosis: a pilot cross-sectional study. J Neurol Sci. 2019 Jan 15;396:87-93. doi: 10.1016/j.jns.2018.11.003. Epub 2018 Nov 3. PMID 30445232
- [Derived] Jimenez-Capdeville ME, Chi-Ahumada E, Garcia-Ortega F, Castanedo-Cazares JP, Norman R, Rodriguez-Leyva I. Nuclear Alpha-Synuclein in Parkinson's Disease and the Malignant Transformation in Melanoma. Neurol Res Int. 2025 Jan 6;2025:1119424. doi: 10.1155/nri/1119424. eCollection 2025. PMID 39816956

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Skin retro auricular biopsies were taken from 67 patients and 20 controls. The biopsies underwent immunohistochemistry (IHC) and immunofluorescence (IF) testing for a-synuclein, after which its presence was quantified as the percentage of positive cells (containing alpha-synuclein). Patients were divided into those with Parkinson's Disease (PD: 34) and those with Atypical Parkinsonism (AP: 33). AP patients included AP with neurodegenerative disease (proteinopathies) and secondary AP
Pre-assignment Details: PD used the United Kingdom PD Society Brain Bank. Lewy body dementia (LBD) used the consortium report on the DLB international workshop.
  AD used the recommendations from the National Institute on Aging and Alzheimer's Association workgroups on diagnostic guidelines for AD.
  MSA used the Second consensus statement on the diagnosis of multiple system atrophy.
  PSP used the report of the NINDS-SPSP International Workshop.
Groups:
- Parkinson Disease: Patients with Parkinson Disease (PD) PD is the patient initially presented asymmetric onset (with both rest and postural tremors with a frequency of between 5 and 7 Hz), rigidity, bradykinesia, postural instability, an acceptable and sustained response to levodopa, and previous and concomitant nonmotor characteristic semiology.
- Atypical Parkinsonism: AP was divided into primary (neurodegenerative) and secondary (postencephalitic, vascular, drug-induced, toxic) groups.
  The neurodegenerative included patients with the diagnosis of Lewy body dementia (LBD) used the consortium report on the DLB international workshop.
  Patients with the diagnosis of AD used the recommendations from the National Institute on Aging and Alzheimer's Association workgroups on diagnostic guidelines for AD.
  Patients with the diagnosis of MSA used the Second consensus statement on the diagnosis of multiple system atrophy.
  The diagnosis PSP used the report of the NINDS-SPSP International Workshop. CBS and we included a case with a diagnosis of neurodegeneration with brain iron accumulation syndrome (NBIA).
  Most of these criteria are summarized in the SIC Task Force appraisal of clinical diagnostic criteria for Parkinsonian disorders.
- Control Group: Subjects apparently in a good state of health without antecedents of neurodegenerative diseases and not symptoms or signs of neurodegeneration (comparable with the group's problem in gender, age, and population characteristics).
Period: Overall Study
Arm/Group | Parkinson Disease | Atypical Parkinsonism | Control Group
Started | 34 | 33 | 20
Completed | 34 | 33 | 20
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Parkinson Disease: Patients with Parkinson Disease: 34 Average. Age (mean SD) 66.82 (+11.4)
- Atypical Parkinsonism: Participants with Atypical Parkinsonism degenerative (26) or secondary (7), total: 33
- Control Group: Subjects without neurodegenerative disease and apparently good state of health (20)
- Total: Total of all reporting groups
Arm/Group | Parkinson Disease | Atypical Parkinsonism | Control Group | Total
Number analyzed (Participants) | 34 | 33 | 20 | 87
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 28 | 26 | 10 | 64
  >=65 years | 6 | 7 | 10 | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.82 (11.4) | 68.2 (13.5) | 74 (7.9) | 69.6 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 11 | 11 | 32
  Male | 24 | 22 | 9 | 55
Region of Enrollment [Count of Participants; unit: Participants]
  Mexico | 34 | 33 | 20 | 87

OUTCOME MEASURES:

1. Primary Outcome: Demonstrate the Presence of Alpha-Synuclein Inclusions in the Skin of Parkinson's Disease and Compare With an Atypical Parkinsonism Group and With a Healthy Control Group.
Description: The presence in the brain of a-synuclein containing Lewy neurites, or bodies, is the histological hallmark of Parkinson's disease (PD).
  The discovery of alpha-synuclein aggregates in nerve endings of the heart, digestive tract, and skin has lent support to the concept of PD as a systemic disease.
  First, our goal was to demonstrate the presence of alpha-synuclein inclusions in the skin of PD patients.
  Second, to detect quantitative differences (measures in the percentage of presence in the skin´s cells) between patients with PD, atypical parkinsonism (AP), compared with an apparent healthy group.
Time Frame: An average of seven days.
Population: PD diagnosis is made if bradykinesia is associated with rigidity, tremor, or postural instability and unilateral onset and persistent asymmetry, excellent response to levodopa, severe levodopa-induced dyskinesia, and progression. AP are other neurodegenerative diseases with parkinsonism or related to strokes, head injuries, encephalitis, neuroleptic use, toxins, cerebral tumor, hydrocephalus. The Control group was a comparable population without parkinsonism and apparently healthy.
Measure: Median (95% Confidence Interval); unit: percentage of expression
Groups:
- Parkinson Disease: Patients with the clinical diagnosis of Parkinson Disease
- Atypical Parkinsonism: Atypical parkinsonian conditions mainly comprise progressive supranuclear palsy (PSP), corticobasal degeneration (CBD), multisystem atrophy (MSA), and dementia with Lewy bodies (DLB). Apart from these sporadic neurodegenerative disorders, atypical parkinsonism has also been described in various other inherited degenerative conditions such as frontotemporal dementia (FTD), Alzheimer's disease, and Perry syndrome. Nondegenerative parkinsonisms include vascular, toxic (use of neuroleptics, exposure to manganese, carbon monoxide, etc.), and traumatic.
- Control Group: Apparently, healthy subjects without a family history of neurodegenerative or chronic diseases could have population characteristics comparable to the problem groups' participants.
Arm/Group | Parkinson Disease | Atypical Parkinsonism | Control Group
Number analyzed (Participants) | 34 | 33 | 20
percentage of expression
  Epidermis. Alpha synuclein expresion | 57.9 [44.9 to 62.6] | 6.9 [0 to 18.3] | 0 [0 to 1.7]
  Pilosebaceus unit | 62.1 [48.5 to 71.2] | 7.7 [0 to 20.7] | 0 [0 to 0]
  Eccrine gland | 58.4 [47.4 to 69.3] | 0 [0 to 0] | 0 [0 to 0]
Statistical Analysis 1: Comparison: Parkinson Disease vs Atypical Parkinsonism vs Control Group; The patients were stratified according to the clinical diagnosis made on the basis of the clinical findings, the MRI, and the progression of the disease. Both the clinical diagnosis and the semiquantitative histological analysis were carried out independently and blind to each other. The presence of aggregates of abnormal a-synuclein, expressed as the percentage of cells with positive inclusions in each experimental group, was tested for normality with the Shapiro-Wilk test; Test type: Superiority — IHC analyses revealed intense α-synuclein positive immunostaining in PD patients, showing small nodular deposits from 1 to 2 μm in diameter in the SCL of the epidermis including the epidermal component adjacent to hair follicles, and in cells from PSUs, while control subjects presented null immunoreaction. The α-synuclein inclusions in the two groups of patients were morphologically similar but quantitatively different. These inclusions appeared to be juxtanuclear; p < 0.01, Kruskal-Wallis — The presence of alpha-synuclein aggregates expressed as % of cells with inclusions was tested for normality (Shapiro-Wilk test). Then, with the nonparametric Kruskal-Wallis followed by Mann-Whitney U tests (software Statistica 7.0 at 95% confidence); The groups were analyzed with Kruskal-Wallis followed by Mann-Whitney U tests; Median Difference (Net) = 57.9, 95% CI 2-sided [44.9 to 62.6], Standard Deviation 8.85 — The expression of the abnormal protein (alpha-synuclein) must be different between the three groups (PD, AP, and control); The patients were stratified according to the clinical diagnosis based on the clinical findings, the MRI, and the progression of the disease. Both the clinical diagnosis and the semiquantitative histological analysis were carried out independently and blind to each other. The presence of aggregates of abnormal α-synuclein, expressed as the percentage of cells with positive inclusions in each experimental group, was tested for normality with the Shapiro-Wilk test. Next, the groups were analyzed with the nonparametric Kruskal-Wallis followed by Mann-Whitney U tests. One independent analysis was performed for each structure, namely the epidermis, PSU, and EG. Assessments were performed using the software Statistica 7.0 (Tulsa, OK) at 95% confidence

ADVERSE EVENTS:
Time Frame: The participants were aware of the possibles adverse events that they could present (pain and bleeding in the site where the biopsy was talked) during the seven days following the biopsy.
Description: Three possible EA were systematically advertised to the patients:
  1. Pain in the retro-auricular area where the biopsy was taken.
  2. Bleeding in the site of the biopsy.
  3. A potential danger of infection in the place of the biopsy. All of them are graduated as AE grade 1, according to the CTCAE. No one event serious event was reported.
Groups:
- PD (n = 34): We enrolled 34 participants who had PD.
- Atypical Parkinsonism (n=33): A total of 33 patients had AP: from they 26 were found to have a neurodegenerative disease clinically (18 had a synucleinopathy-related diagnosis: MSA, LBD, and 8 had tauopathies: PSP, AD). We also included seven patients with secondary parkinsonism.
- Control Group (n=20): A control group (n = 20) of similar age and sex distribution to the patient population was included. There was no significant difference in either age or evolution of disease between the two groups with parkinsonism.
Arm/Group | PD (n = 34) | Atypical Parkinsonism (n=33) | Control Group (n=20)
All-Cause Mortality (participants affected / at risk) | 0/34 | 0/33 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/33 | 0/20
Other Adverse Events (participants affected / at risk) | 1/34 | 1/33 | 0/20
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | PD (n = 34) (N=34) | Atypical Parkinsonism (n=33) (N=33) | Control Group (n=20) (N=20)
Transient bleeding (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 — Transient bleeding that stops with local biopsy site compression.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No